CLINICAL TRIAL: NCT01934374
Title: Long-Term Effects of Task-Oriented Lower Extremity Strengthening Training on Functional Connectivity of the Brain, Motor Functions, Physical Activity Level, and Quality of Life in Patients With Subacute Stroke
Brief Title: Long-Term Effects of Task-Oriented Lower Extremity Strengthening Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 200812148R
Record Dates: First submitted 2013-08-08; First posted 2013-09-04 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-08

CONDITIONS: Ischemic Cerebrovascular Accident
Keywords: task-oriented training, long-term effects, plasticity
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stroke (Experimental): On the 30th day post stroke (D30), the exjperimental group will start to receive the task-oriented lower extremity strengthening training (TOLEST) program for four weeks, one hour per session and three sessions per week. The TOLEST focuses on using task-specific circuit training combined with strengthening of bilateral lower limbs.
  Interventions: Behavioral: Task-Oriented Lower Extremity Strengthening Training
- Control (No Intervention): The control group will receive equal-dose exercises starting on D30, with the emphasis on stretching and non-functional movements of the affected lower extremity.

INTERVENTIONS:
Behavioral: Task-Oriented Lower Extremity Strengthening Training — On the 30th day post stroke (D30), the experimental group will start to receive the TOLEST program for four weeks, one hour per session and three sessions per week. The TOLEST focuses on using task-specific circuit training combined with strengthening of bilateral lower limbs.
  The control group will receive equal-dose exercises starting on D30, with the emphasis on stretching and non-functional movements of the affected lower extremity.
  Arms: Stroke

SUMMARY:
Task-oriented exercises combined with strengthening have been shown effective in improving walking functions in patients with chronic stroke. However, similar approaches of therapeutic exercises have not been applied to subacute stroke with long-term follow-up, using outcome measures across the three levels of functioning (body functions/structure, activities, and participation) of the International Classification of Functioning, Disability, and

Health (ICF) model. Therefore, this study will be conducted to fulfill three purposes:

1. To investigate the long-term effects of a four-week task-oriented lower extremity strengthening training (TOLEST) program in patients with subacute stroke;
2. To investigate the interrelationships among functional connectivity of the brain, lower extremity motor functions, physical activity level, and quality of life in patients with stroke who have received this four-week TOLEST program in the subacute phase of stroke; and
3. To identify prognostic factors for recovery in functional connectivity of the brain, lower extremity motor functions, physical activity level, and quality of life in patients with stroke who have received this four-week TOLEST program in the subacute phase of stroke.

DETAILED DESCRIPTION:
We conducted a meta-analysis to examine the effects of task-oriented approach in patients with sub-acute stroke and a preliminary study of an assessor-blind randomized controlled trial with a total of 3 patients with sub-acute stroke (experimental group: E1; control group: C1 and C2). The participants were randomly assigned to the experimental group or the control group. All participants received 4 weeks of exercise training, which were 4 sessions per week and 60 minutes for each session. The experimental group received task-oriented circuit training to improve lower extremity motor functions. The control group received stretch exercises and upper extremity activities in sitting posture. Both groups received clinical asessments on lower extremity motor functions (primary outcomes), the structural integrity of the CST using diffusion spectrum imaging, and the cortical activation patterns of the SMC using functional magnetic resonance imaging(secondary outcomes) at baseline, post-training (week 4), and 1 month follow-up (week 8). Because of the small number of subjects, we also included one subject (E2) who received the same training programs as experimental group in our pilot study as one subject of the training group result. Training effects were descriptively analyzed for individual subjects.

The meta-analysis results showed that task-oriented training led to significantly greater improvement than other training on 6-minute walking distance (mean difference = 82.49 meter; 95% confidence interval: 27.59-137.38) and comfortable gait speed (standardized mean difference = 0.27; 95% confidence interval: 0.03-0.52) in patients with subacute stroke. Our preliminary results showed that the experimental group achieved meaningful improvements in most of the primary outcomes but not for the control group. In addition, different brain reorganization patterns were observed in the two groups.

The results of meta-analysis provide relevant clinical evidence for the effects of task-oriented training on lower extremity motor functions, and this preliminary study provides the pilot result for the effects of task-oriented circuit training on lower extremity motor functions, brain structural and functional plasticity in patients with sub-acute stroke.

ELIGIBILITY:
Inclusion Criteria:

1. in the subacute stage of stroke (within 20 to 30 days post-onset) and stable medical condition;
2. presence of residual gait impairment;
3. being able to walk 5 m with or without assistive device independently;
4. the paretic lower leg being able to perform at least 10 degrees of active ankle dorsiflexion from the resting position;
5. no apparent spasticity in affected leg to interfere the affected limb movement (Modified Ashworth Scale < 2)

Exclusion Criteria:

1. claustrophobia and indwelling metals or implanted devices incompatible with fMRI testing;
2. serious cardiac conditions (e.g. unstable angina serious cardiac arrhythmias, heart failure, hypertrophic cardiomyopathy, severe aortic stenosis, pulmonary embolus, or infarction);
3. symptoms or history of other neurological or orthopedic problems which would affect their lower limb function;
4. severe cognitive, perceptual, or communication problems

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
10-meter walk test | up to 4 weeks, change from baseline to 4 weeks

SECONDARY OUTCOMES:
Functional MRI (fMRI), diffusion spectrum imaging (DSI) | up to 4 weeks, change from baseline to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Fang Tang, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Pei-Fang Tang, Taipei, Taiwan, Taiwan